CLINICAL TRIAL: NCT00347204
Title: Double Masked Evaluation of Acular LS Versus Nevanac for Postoperative Pain Control in Eyes Undergoing PRK
Brief Title: Comparison of Acular LS Versus Nevanac for Pain Control in Eyes Undergoing PRK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center For Excellence In Eye Care (Other)
Collaborators: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5225; NCT00405028 (obsolete NCT alias)
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Myopia; Hyperopia
Keywords: PRK; laser vision correction; surface ablation; pain; wound healing; corneal haze
MeSH Terms: conditions — Myopia; Hyperopia; Pain; Corneal Opacity | interventions — Ketorolac; nepafenac

INTERVENTIONS:
Drug: ketorolac (Acular LS)
Drug: Nepafenac (Nevanac)

SUMMARY:
To determine the ability of two topical Nonsteroidal Anti-inflammatory drops (Acular LS & Nevanac) to help control pain following Photorefractive Keratectomy (PRK).

DETAILED DESCRIPTION:
Laser Vision Correction is the most commonly performed elective surgical procedure in the United States. Although Laser-Assisted in-situ Keratomileusis (LASIK) is the more popular technique, a growing number of surgeons have switched to surface ablation techniques, including PRK, LASEK and Epi-LASIK.1 With surface laser procedures, the corneal epithelium is removed by a variety of techniques (laser, manual debridement, diluted alcohol2,3, epi-keatome) prior to laser reshaping of the corneal stroma. Following the procedure, a contact lens is placed on the eye to promote epithelial regeneration. Due to the size of the epithelial defect, it can take between 3 to 6 days for the epithelium to regenerate. During this healing process, patients often complain of moderate to severe ocular pain, and delayed healing may result in an increased risk of infection or corneal haze4.

Over the past decade, a variety of methods have been used to assist with reducing pain following surface laser procedures. Topical Nonsteroidals have been shown in a number of studies to help reduce the degree of pain following PRK. Topical dilute tetracaine has also been shown to assist with the reduction of pain following PRK. Oral pain medications, such as Vioxx, Celebrex, and even Prednisone have been recommended as additional treatment options for pain control.

In October 2005, a new topical nonsteroidal anti-inflammatory drop, Nevanac, was approved by the FDA. Nevanac was approved with a a TID dosing schedule.

Acular LS is the current market leader for topical NSAID eye drops. Acular LS is typically used on a QID dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PRK for myopia or hyperopia

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-01; Study Completion 2006-06

PRIMARY OUTCOMES:
Prevention of postoperative discomfort on postoperative days 1 to 5 after PRK
Best-corrected Visual acuity at all study visits
Degree of corneal haze at all study visits
Time to epithelial closure in each eye after PRK

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Principal Investigator — Center For Excellence In Eye Care